# **HPV Vaccine to Interrupt Progression of Vulvar and Anal Neoplasia (VIVA)**

Trial: A Randomized, Double-Blind, Placebo-Controlled Trial

**Study Protocol** 

Version 12.0 14 December 2021 Principal Investigators: Margaret M. Madeleine, PhD

Fred Hutchinson Cancer Research Center 1100 Fairview Ave N., PO Box 19024

Seattle, WA 98109

Telephone: (206) 667-4629 Email: mmadelei@fhcrc.org

Anna Wald, MD, MPH, University of Washington

Harborview Medical Center, 325 9<sup>th</sup> Ave Virology Research Clinic, Box 359928

Seattle, WA 98104

Telephone: (206) 520-4340 Email: <a href="mailto:annawald@uw.edu">annawald@uw.edu</a>

Clinical Co-Investigators: Constance Mao, MD

Jeffrey Schouten, MD Verena Grieco, MD

Helen Stankiewicz Karita, MD

Warner Huh, MD
Maggie Liang, MD
Haller Smith, MD
Kerri Bevis, MD
Charles Leath, MD
J. Michael Straughn, MD
Rebecca Arend, MD

**Statistician:** Amalia Magaret, PhD, University of Washington

Harborview Medical Center, 325 9<sup>th</sup> Ave Virology Research Clinic, Box 359928

Seattle, WA 98104

Study Sites: University of Washington Virology Research Clinic

908 Jefferson St. Suite 11NJ-1166 Seattle, WA 98104

University of Alabama at Birmingham

1700 6<sup>th</sup> Ave. So., 176F Bldg Birmingham, AL 35233

# **TABLE OF CONTENTS**

| PRC | OTOCOL SUMMARY | 6 |
|-----|-------------------------------------------|----|
| GLC | OSSARY OF TERMS | |
| LIS | T OF ABBREVIATIONS | 9 |
| 1 | BACKGROUND | 11 |
| 1 | .1 Burden of Disease | 11 |
| | .2 PRIOR EVIDENCE OF SAFETY | |
| 2 | HYPOTHESIS, STUDY OBJECTIVE, AND OUTCOMES | |
| | .1 HYPOTHESIS | |
| | .3 OUTCOMES | |
| | 2.3.1 Primary Endpoint | |
| | 2.3.2 Secondary Endpoints | |
| 3 | STUDY DESIGN | 12 |
| 4 | PARTICIPANT SELECTION | 13 |
| 1 | .1 Inclusion Criteria | 15 |
| | .2 EXCLUSION CRITERIA | |
| | .3 RECRUITMENT PROCESS | |
| 5 | STUDY PROCEDURES | 14 |
| 5. | .1 SCREENING VISIT (VISIT -1) | 14 |
| | .2 ENROLLMENT VISIT (MONTH 0) | |
| | .3 Months 2 and 6 | |
| | .4 Month 7 | |
| | .5 MONTHS 18, 24, AND 36 | |
| | .6 MONTHS 12 AND 42 | |
| | .8 DUAL SITE LESIONS | |
| | .9 RANDOMIZATION AND BLINDING | |
| | .10 REMOTE CONSENTING | |
| 5. | .11 UNBLINDING PARTICIPANTS | 18 |
| 6 | POTENTIAL RISKS & BENEFITS | 19 |
| | .1 POTENTIAL RISKS | 19 |
| 6. | .2 POTENTIAL BENEFITS | 20 |
| 7 | CLINICAL PROCEDURES | 20 |
| | .1 BLOOD COLLECTION | |
| | .2 HPV SWAB COLLECTION | |
| | .3 HPV ORAL RINSE COLLECTION | |
| | .4 DATA COLLECTION | |
| | .6 ANAL BIOPSY | |
| | .7 Vulvoscopy | |
| 7. | .8 VULVAR BIOPSY | 22 |
| 8 | LABORATORY PROCEDURES | 22 |
| 8. | .1 URINE PREGNANCY TESTING | 22 |

| | 8.2 | HIV-1 Antibody Testing | |
|----|--------------|-------------------------------------------|----|
| | 8.3 | HPV Capsid Antibody Analysis | 23 |
| | 8.4 | HPV TYPING FROM TISSUE | |
| | 8.5 | HPV TYPING FROM ORAL SAMPLES | 23 |
| | 8.6 | FUTURE GENETIC RESEARCH | 23 |
| 9 | STU | JDY PRODUCT | 23 |
| | 9.1 | TREATMENT GROUPS | 23 |
| | 9.2 | STUDY PRODUCT AND SOURCE | 23 |
| | 9.3 | STORAGE | |
| | 9.4 | RECOMMENDED DOSE AND SCHEDULE | |
| | 9.5 | ADMINISTRATION | |
| | 9.6 | CONTRAINDICATIONS | |
| | 9.7 | BLINDING | |
| | 9.8 | STUDY PRODUCT ACCOUNTABILITY | |
| 10 | ) A | ASSESSMENT OF SAFETY | 25 |
| | 10.1 | ADVERSE EVENTS | |
| | 10.2 | DEFINITION OF ADVERSE EVENT | |
| | 10.3 | DEFINITION OF SERIOUS ADVERSE EVENT (SAE) | |
| | 10.4 | ADVERSE EVENT REPORTING | |
| | 10.4 | , g | |
| | 10.4<br>10.5 | , | |
| | | 5.1 Data and Safety Monitoring Plan | |
| | | 5.2 Data and Safety Monitoring Plan5.2 | |
| | | , , | |
| 11 | | CLINICAL MANAGEMENT | |
| | 11.1 | PARTICIPANT WITHDRAWAL OR DISCONTINUATION | 28 |
| 12 | 2 [ | DATA MANAGEMENT | 29 |
| | 12.1 | DATA COLLECTION | 29 |
| | 12.2 | CASE REPORT FORMS (CRF) | 29 |
| 13 | 3 F | IUMAN SUBJECTS PROTECTIONS | 29 |
| | 13.1 | IRB Approval | 29 |
| | 13.2 | INFORMED CONSENT | |
| | 13.3 | PROTECTION AGAINST RISK | 30 |
| 14 | 4 S | STUDY DESIGN DETAILS | 30 |
| | 14.1 | SAMPLE SIZE | 30 |
| | 14.2 | RANDOMIZATION | |
| 1 | 5 S | STATISTICAL CONSIDERATIONS | 31 |
| | 15.1 | MISSING DATA AND LOSS TO FOLLOW-UP | 31 |
| | 15.2 | VISIT WINDOWS | |
| 16 | 6 S | STATISTICAL ANALYSIS PLAN | 31 |
| | 16.1 | Data handling | 21 |
| | 16.2 | ANALYSIS POPULATIONS | |
| | 16.3 | PRIMARY ENDPOINT | |
| | 16.4 | SECONDARY ENDPOINTS | |
| | | DEPARTURES FROM MODEL ASSUMPTIONS | |

| 16.6 | LEFT TRUNCATION | .33 |
|--------|----------------------------|------|
| 17 F | REFERENCES | . 34 |
| APPENI | DIX A: STUDY VISIT WINDOWS | . 36 |
| ΔΡΡΕΝΙ | DIX B. TABLE OF PROCEDURES | 37 |

## PROTOCOL SUMMARY

**Design**: Randomized, double-blind, placebo-controlled clinical trial

**Population**: Participants with anal (men and women with AIN2/3) or vulvar (women

with VIN2/3) high-grade squamous intraepithelial lesions (HSIL)

**Aim**: To compare persistent high-risk HPV infection rates (by PCR detection of

the same high-risk HPV vaccine type in ≥ 2 consecutive samples) among

vaccine compared with placebo recipients

**Sub-Aims:** 1) To measure time to subsequent HSIL among vaccine compared to

placebo recipients

2) To investigate the role of natural antibodies in deterring persistent infection among placebo recipients and magnitude of vaccine antibody among those who did and did not have a persistent infection in the

vaccine recipients

3) To compare persistent high-risk HPV oral infection rates among

vaccine compared with placebo recipients

Sample Size: 230 participants

**Study Sites**: University of Washington

Virology Research Clinic

Seattle, WA

University of Alabama at Birmingham

Gynecologic Oncology Clinic

Birmingham, AL

Study Duration: Clinic visits through Month 36 and telephone follow-up through Month 42

We will conduct a randomized, double-blind, placebo-controlled, proof-of-concept clinical trial of Gardasil, a 9-valent HPV vaccine (**9vHPV**), administered as treatment for anal or vulvar HSIL after initial treatment. We will enroll 230 individuals with anal or vulvar HSIL, identified from the local SEER cancer registry or by physician referral. Participants will be randomized 1:1 to vaccine or placebo. This study will take place at the University of Washington (**UW**) Virology Research Clinic (**VRC**) and at the University of Alabama at Birmingham (**UAB**) Gynecologic Oncology Clinic. The Screening Visit includes consent forms, an HIV test, review of the eligibility criteria, colposcopy (vulvoscopy for those with prior vulvar HSIL and anoscopy for those with prior anal HSIL) with a biopsy if clinically indicated, swab sample of colposcopy site, and oral rinse for HPV DNA detection. Eligible participants will return for an Enrollment Visit in which they will undergo a blood draw, baseline questionnaire, and then be randomized to receive the vaccine or placebo (at 0, 2, and 6 months). Follow-up visits will occur at Months 7, 18, 24, and 36. Procedures at follow-up visits include a blood draw and oral rinse at Month 7; a blood draw, oral rinse, and anoscopy/vulvoscopy for surveillance at Months 18 and 36; and an oral rinse and swabs of the qualifying lesion site at Month 24. Telephone or web-based interviews will be

conducted at Months 12 and 42. Participants will receive an anoscopy or vulvoscopy at Months 0, 18, and 36, with biopsies as needed if a lesion is visualized at the Month 0,18, and 36 visits. Slides from tissue samples for the qualifying lesion and potential HSIL recurrence lesions collected during follow up will be evaluated centrally by the study pathologist. We hypothesize that the vaccine will reduce risk of high-risk HPV type-specific persistence of vaccine types by 50%.

## **GLOSSARY OF TERMS**

| Low grade squamous intraepithelial neoplasia (LSIL) | Based on the Lower Anogenital Squamous Terminology (LAST project), LSIL includes the following: • HPV effect (condyloma, koilocytosis) • Mild dysplasia • VIN1 /AIN1 These diagnostic terms are used to reference the same underlying condition. |
|---|---|
| High grade squamous intraepithelial neoplasia (HSIL) | Based on the LAST project, HSIL includes the following: • Moderate dysplasia • VIN2 or AIN2, with p16 staining as needed to rule out low-grade disease • Severe dysplasia • Carcinoma in situ • VIN3 or AIN3 These diagnostic terms are used to reference the same underlying condition. |
| Single site | Participant with history of histologically confirmed initial or recurrent anal HSIL or vulvar HSIL either on or after 1/1/2014. |
| Dual sites | Participant with a history of histologically confirmed initial or recurrent anal and vulvar HSIL (both sites), with at least one HSIL diagnosed on or after 1/1/2014 |
| Study inclusion criteria in participants with history of HSIL at <b>single site</b> | Study eligibility is based on having an anal or vulvar HSIL lesion (initial or recurrence) either on or after 1/1/2014. |
| Study inclusion criteria in participants with history of HSIL at <b>dual sites</b> | Participants with history of HSIL at both sites will have only one site included in the main analysis: |
| | most recently treated; or |

| | <ul> <li>2) if both treated at the same time, the lesion diagnosed closest to 1/1/2014; or</li> <li>3) if both treated and diagnosed at the same times, flip a coin.</li> </ul> |
|---|---|
| Qualifying lesion | Histopathologically confirmed anal or vulvar HSIL diagnosed closest to (on or after) 1/1/2014 |
| Criteria for randomization | Randomization criteria: 1) Anatomic site (vulvar or anal) 2) HIV status (positive or negative) 3) <b>Time since diagnosis</b> of the qualifying lesion (< 12 months or > 12 months) |
| Persistent Infection | PCR detection of the same high-risk HPV vaccine type in ≥ 2 consecutive samples |

#### LIST OF ABBREVIATIONS

AAHS amorphous aluminum hydroxyphosphate sulfate

AE adverse event

AIN2 anal intraepithelial neoplasia grade 2
AIN3 anal intraepithelial neoplasia grade 3

ANCHOR anal intraepithelial neoplasia grades 2 (p16+) or 3; anal HSIL

ANCHOR Anal Cancer HSIL Outcomes Research Study (NCT02135419)

cc cubic centimeter

CDC Centers for Disease Control

CIN2/3 cervical intraepithelial neoplasia grades 2 and 3

CRF case report forms

CROI Conference on retroviruses and opportunistic infections

CRS clinical research support

CSS Cancer Surveillance System, the SEER cancer registry for the

**Puget Sound Region** 

CTCAE common terminology criteria for adverse events

DSMB Data Safety Monitoring Board

DSMC Data and Safety Monitoring Committee

FDA Food And Drug Administration

FHCRC Fred Hutch Cancer Research Center

HIPAA Health Insurance Portability And Accountability Act

HIV human immunodeficiency virus

HPV human papillomavirus
HRA high resolution anoscopy
HSD Human Subjects Division

HSIL high-grade squamous intraepithelial lesion

ID identification data

IRB Institutional Review Board ITT intention to treat analysis

mcg Microgram

NCT National Clinical Trial

PCR polymerase chain reaction

PE physical exam

PHI protected health information

PP per protocol analysis

RCT randomized controlled trial

SAE serious adverse event

SEER Surveillance, Epidemiology, and End Results Program

SOP Standard Operating Procedures

SRC Scientific Review Committee

UW University of Washington

VIN2 vulvar intraepithelial neoplasia grade 2

VIN2/3 vulvar intraepithelial neoplasia grade 2 or 3; vulvar HSIL

VIVA Vaccine to Interrupt progression of Vulvar and Anal neoplasia trial

NCT03051516

VLP virus like particle

VRC Virology Research Clinic

°C degrees centigrade

4vHPV quadrivalent human papillomavirus vaccine
9VHP nonavalent human papillomavirus vaccine

#### 1 BACKGROUND

#### 1.1 Burden of Disease

In the U.S., over 10,000 cases of anal and vulvar cancer are diagnosed annually, and most are HPV related.<sup>1</sup> Although mortality from anal and vulvar HSIL is low, there is a high rate of recurrence: approximately 30% recur within 5 years with higher recurrence in HIV-infected individuals.<sup>2</sup> Development of recurrence(s) necessitates repeated surgeries associated with reduced function.<sup>3</sup> We estimate a prevalence of nearly 90,000 individuals with anal or vulvar HSIL among those diagnosed in the last 10 years in the US; in addition, the number of incident cases is increasing annually at a gradual but steady rate. As the unvaccinated population ages, HSIL will also continue to increase.

We propose to conduct a randomized, double-blinded, placebo-controlled clinical trial to evaluate whether the risk of recurrence of HSIL can be reduced by vaccination with 9vHPV. These lesions have the highest likelihood of HPV-related anogenital pre-cancers to progress to cancer, are more likely than invasive lesions to respond to the vaccine, and over 90% are caused by HPV types contained in the 9vHPV vaccine.<sup>1, 4</sup>

This trial will be among the first to measure the potential benefit of the vaccine as an adjunct to treatment for HSIL, and the first to include non-HIV seropositive individuals and women with VIN2/3. Prior studies of prophylactic HPV vaccine efficacy avoided enrolling HPV positive individuals, and attempts to pool information from the small numbers of HPV positive participants enrolled in those trials suffer from heterogeneity due to different designs, goals, and outcomes of the pooled studies. Two observational studies have compared outcomes among vaccinated and unvaccinated individuals with HPV-related cancer, 6, 7 and three randomized trials of HPV-related lesion recurrence are currently recruiting. In South Africa, a randomized trial will assess the impact of 4vHPV vaccine against recurrence of CIN2/3 (NCT01928225) among 180 HIV+ women followed for 1 year, which may limit the number of events detected. Another RCT (NCT02087384), is being conducted at 4 centers in the Netherlands, and will assess 4vHPV against anal HSIL recurrence among HIV positive MSM. In a third trial within the AIDS Malignancy Consortium (NCT01461096), 464 HIV-infected MSM will be randomized to 4vHPV and followed for 3 years. These complementary trials are conducted exclusively in HIV positive individuals. We anticipate that approximately 70% of trial participants in the VIVA Trial will be HIV negative. Our target population will be primarily identified from a population-based SEER registry, and advances beyond currently ongoing trials by including HIV negative individuals and women with anal or vulvar HSIL.

Emerging data suggest that the licensed vaccine could decrease risk of recurrence of HSIL by 50%, by increasing immune response and reducing the risk of reactivation of disease. However, a recent HPV trial in HIV infected individuals with no previous HPV-associated cancers was stopped early due to lack of difference between the placebo and vaccine arms with regard to prevention of new HPV infections or to improve treatment outcomes. As this study was stopped early, follow-up time was limited to assess anal HSIL risk. We recognize that the most effective use of the vaccine is before sexual debut; this is very clear. However, the potential benefits of the vaccine are to reduce recurrence of HSIL and avoid multiple and increasingly disfiguring surgeries, psychosexual trauma, and debilitated functions through relatively low cost and, as we hope to prove, safe vaccination.

The WHO has recommended high-risk HPV persistent infection be evaluated as an intermediate endpoint for HPV vaccine efficacy. <sup>9, 10</sup> Persistence is generally defined as the same HPV type identified at consecutive time points. <sup>11, 12</sup> This virologic approach to the primary aim is associated with a higher frequency of outcomes and therefore allows us to reduce the sample size to 230 people. However, this change also comes with the limitation that we may detect persistent infections that do not develop into histologic HSIL recurrence. Given these

considerations, the original primary aim, time to recurrence of HSIL, will become a secondary aim.

## 1.2 Prior Evidence of Safety

The common reported adverse events from the licensure for 9-valent HPV vaccine trials<sup>13, 14</sup> report injection site reaction and lightheadedness, likely resulting from pain of injection. No clinically important safety concerns have emerged from those studies or studies during implementation.<sup>15-17</sup> Safety of the vaccine after treatment for HSIL is unknown, but the vaccine is likely to be safe in that population. As our study will result in off-label use, we will monitor safety by comparing type and frequency of AEs in the two study arms.

## 2 HYPOTHESIS, STUDY OBJECTIVE, AND OUTCOMES

## 2.1 Hypothesis

The main purpose of this trial is to test whether an FDA approved prophylactic HPV vaccine (9vHPV) will lead to a 50% reduction of persistent HPV compared to unvaccinated individuals with HSIL.

## 2.2 Study Objective

We will test if the 9vHPV vaccine delivered after treatment for HSIL reduces the risk of persistent high-risk infection by 50% in the vaccinated *vs.* placebo arms. We will also evaluate safety of the HPV vaccine in HSIL participants.

#### 2.3 Outcomes

## 2.3.1 **Primary Endpoint**

The primary endpoint of the study is time to persistent high-risk infection among vaccine compared with placebo recipients.

## 2.3.2 **Secondary Endpoints**

We will assess the safety of the vaccine.

We will additionally evaluate vaccine efficacy against recurrence after adjustment for baseline stratification variables. The impact of HPV antibody level on persistence and recurrence will be evaluated separately by vaccination arm.

#### 3 STUDY DESIGN

We will conduct a randomized, double-blind, placebo-controlled proof-of-concept clinical trial of 9vHPV administered as an adjunctive treatment for anal or vulvar HSIL. We will enroll 230 individuals, identified using either the local SEER cancer registry, to which individuals with HSIL (AIN3/VIN3) are reported, or physician referral of participants with HSIL (AIN2/VIN2) that are confirmed by a pathologist. This study will be conducted at the research clinics, where all procedures and specimen collection will be performed by experienced research clinicians. The

7-8 clinic visits include a screening visit, three vaccination visits (at 0, 2, and 6 months), and four follow up visits (at 7, 18, 24, and 36 months). Phone call follow-ups will take place at months 12 and 42 months. In some participants, the screening and the enrollment visit may be combined.

#### 4 PARTICIPANT SELECTION

#### 4.1 Inclusion Criteria

Men and women who meet all the following criteria are eligible for inclusion in this study:

- Age 27- 69 at enrollment
- Histologically confirmed diagnosis of initial or recurrent anal or vulvar high-grade squamous intraepithelial lesion (AIN2/3 or VIN2/3) diagnosed on or after 1/1/2014; study pathologist will use p16 staining as needed to rule out LSIL disease
- > 2 months since last therapy for HSIL.
- No clinical evidence of HSIL on screening examination; if HSIL is suspected, a biopsy will be done to exclude HSIL. Patients whose screening visit reveals HSIL on biopsy, may be re-screened  $\geq 2$  months after therapy.
- Resident in the catchment area of the clinics willing to attend up to 8 clinic visits for a 36-month period
- Sexually active women of child-bearing potential must be willing to use effective contraception through Month 7 of the study
- If HIV positive, receipt of anti-retroviral therapy continuously for at least 6 months prior to enrollment
- Ability to give informed consent
- Willingness to sign medical records release form and tissue release form

#### 4.2 Exclusion Criteria

Men and women who meet any of the following criteria are not eligible for this study:

- Currently pregnant
- Chemotherapy (current, within the last month, or anticipated in the next 7 months)
- Prior history of invasive HPV-related anogenital cancer (cervical, vaginal, vulvar, penile, or anal cancer), or oropharyngeal cancer (base of tongue, tonsil). Prior cancer at other sites (including most of oral cavity) or larynx are not exclusions
- Unstable medical condition (e.g., another malignancy requiring treatment, malignant hypertension, poorly controlled diabetes, another cancer except for fully excised non-melanoma skin cancer)
- Prior HPV vaccination
- Known allergy or intolerance to lidocaine
- Currently participating in an interventional research study related to HPV, except the ANCHOR study (NCT02135419)
- Any other condition which, in the opinion of the investigator, may compromise the subject's ability to follow study procedures and safely complete the study.

## 4.3 Recruitment Process

We will recruit 230 men and women with prior HSIL and no evidence of current HSIL. Potentially eligible participants will be referred to study staff who will discuss the study and eligibility criteria with the participant. Those that are eligible and interested will arrange a screening appointment at the clinic.

Sources of potential participants include but are not limited to:

- The Cancer Surveillance System (CSS) of the Fred Hutchinson Cancer Research Center, a population-based National Cancer Institute Surveillance, Epidemiology, and End-Results (SEER) cancer registry.
- Physicians referrals
- Pathology records from nearby medical institutions in Seattle and Birmingham
- Community recruitment

All recruitment methods and materials will be IRB approved prior to use.

We will obtain a partial waiver of HIPAA authorization and partial waiver of consent for recruitment.

## 5 STUDY PROCEDURES

## 5.1 Screening Visit (Visit -1)

After receipt of the approach letter or a brochure from their healthcare provider, interested potential participants will be screened by telephone regarding study eligibility criteria. Potentially eligible participants will schedule a Screening Visit.

During the Screening Visit, study background and procedures will be explained. Potential participants will have a chance to ask questions about all aspects of the study. Written informed consent, HIPAA Authorization, and Medical Records and Tissue Releases will be obtained prior to participation in the study. Inclusion/exclusion criteria will be reviewed and the qualifying lesion for inclusion and randomization will be determined:

| Study inclusion in participants with history of HSIL at single site | Study eligibility is based on having a history of an anal or vulvar HSIL lesion (initial or recurrence) either on or after 1/1/2014 and no HSIL at screening. |
|---|---|
| Study inclusion in participants with history of HSIL at <b>dual sites</b> | Participants with history of HSIL at both sites will have only one site included in the main analysis: 1) most recently treated; or 2) if both treated at the same time, the lesion diagnosed closest to 1/1/2014; or 3) if both treated and diagnosed at the same times, flip a coin. |

Demographic and baseline medical history information will be obtained which will include questions about general health, medical conditions, concomitant medications, and anogenital pathology including treatments. Sexually active women of childbearing potential will undergo a urine pregnancy test. Blood will be drawn for HIV testing, if needed. An oral rinse will be collected for HPV DNA detection. A general physical exam will be performed. Anoscopy or vulvoscopy will be performed of the anus or vulva, depending on the location of the qualifying lesion. Swab samples will be collected. A biopsy will be taken if any lesions suspicious for HSIL are visualized at the qualifying site.

If a biopsy is collected during the Screening Visit:

- Participants with negative biopsy results will be eligible for enrollment into the study.
- Participants with HSIL (AIN2/3 or VIN2/3) positive biopsy results will be deferred but will be offered the ability to rescreen ≥2 months after treatment. The results of the anoscopy/vulvoscopy and exam will be shared with the participant and their healthcare provider. Any follow-up treatment will be provided by the outside provider, not by the study.

Individuals who are eligible to enroll in the VIVA Trial at the Screening Visit may undergo a combined Screening Visit and Enrollment Visit. Individuals in need of medical documentation before becoming eligible (i.e., negative HSIL biopsy results or confirmation of HIV status) will be asked to schedule their Enrollment Visit within 8 weeks of their Screening Visit.

Individuals who had anoscopy or vulvoscopy performed within 8 weeks of the Screening Visit by clinical co-investigators or an ANCHOR-certified provider and had no evidence of vulvar or anal HSIL will not need anoscopy or vulvoscopy performed at the Screening Visit. They will undergo all other screening procedures. Documentation of the high resolution anoscopy or vulvoscopy procedure, and any biopsies performed will be requested and reviewed prior to entry to verify that no HSIL was detected on recent HRA or vulvoscopy exams.

## 5.2 Enrollment Visit (Month 0)

Inclusion/exclusion criteria will be reviewed. Interim medical history and concomitant medications will be collected. A targeted physical exam will be performed. Vital signs (blood pressure, pulse, temperature) including self-reported height and weight will be collected. Women of childbearing potential will undergo a urine pregnancy test. Up to 20 cc of blood will be drawn for HPV antibody assays.

Participants will be randomized and the study product will be administered via intramuscular injection in the deltoid region of the preferred arm. Participants will be observed for 15 minutes after vaccine dose administration. Participants will be instructed about potential adverse events (AEs), and provided with a log to record any fever or injection site reactions for the next 5 days.

Participants will complete a self-administered questionnaire.

#### 5.3 **Months 2 and 6**

Interim medical history and concomitant medications will be obtained including any new anogenital biopsies or treatments. A targeted physical exam will be performed. Vital signs (blood pressure, pulse, temperature) will be collected. Women of childbearing potential will undergo a urine pregnancy test prior to each vaccination.

The study product will be administered via intramuscular injection in the deltoid region of the preferred arm. Participants will be observed for 15 minutes after vaccine dose administration. Participants will be instructed about potential AEs, and provided with a log book to record any fever or injection site reactions over the next 5 days.

Participants will complete a self-administered questionnaire at Month 6.

#### 5.4 **Month 7**

Interim medical history and concomitant medications will be obtained including any new anogenital biopsies or treatments. A targeted physical exam will be performed. An oral rinse will be collected for HPV DNA detection. Blood will be drawn (up to 30 cc serum) for HPV antibody assays and DNA (optional).

# 5.5 **Months 18, 24, and 36**

At months 18 and 36, interim medical history and concomitant medications will be obtained including new anogenital biopsies or treatments. A targeted physical exam will be performed. Blood will be drawn (up to 20 cc serum) for HPV antibody assays. An oral rinse for HPV DNA detection will be collected. Swabs will be obtained at the qualifying lesion site of the vulva or anus. Anoscopy or vulvoscopy will be conducted as surveillance for recurrence and a biopsy will be taken of any visible lesion suspicious for HSIL. At Month 36, if a lesion is identified, a biopsy will be taken. If no lesion is identified at Month 36, participants will undergo an optional biopsy at the site of the qualifying lesion. The results of the anoscopy/vulvoscopy and exam will be shared with the participant and their healthcare provider. Any follow-up treatment will be provided by the outside provider, not by the study.

Participants who had anoscopy or vulvoscopy performed within the Months 18 and/or 36 visit windows by a clinical co-investigator or an ANCHOR-certified provider will not need an anoscopy or vulvoscopy performed at the Months 18 and/or 36 Visits. Pathology reports from any biopsies obtained during these exams will be requested and reviewed. Additionally, tissue blocks will be requested for further testing. Participants will undergo all other Month 18 and 36 visit procedures.

Participants will complete a self-administered questionnaire at each of these visits.

At month 24, swabs of the qualifying lesion site and an oral rinse for HPV detection will be obtained.

# 5.6 **Months 12 and 42**

Telephone interviews will be conducted at Months 12 and 42. These short interviews will include questions about health (including any SAEs), smoking status, and anogenital disease.

During the Month 42 telephone interview, participants will now be offered the opportunity to receive their randomization assignment (See section 5.11).

## 5.7 Reminder Calls

Reminder calls will be conducted every 1-3 months after the Month 12 visit for study retention. Reminders will be made by phone, email or text per participant preference.

#### 5.8 **Dual Site Lesions**

Definition of Dual Lesions: Participant with a history of histologically confirmed initial or recurrent anal and vulvar HSIL (both sites), with at least one HSIL diagnosed on or after 1/1/2014.

A complementary HRA or vulvoscopy exam will be offered to individuals with lesions at dual sites or to persons who, in the opinion of the investigators, may benefit from the complementary exam. The complementary HRA or vulvoscopy can be performed at any time after participant enrollment based on participant and clinician availability.

Information about the dual site lesion history will be captured and become part of the study record. Subsequent vulvoscopy or anoscopy will be offered at 18 and 36 months, according to the single site follow up examinations.

## 5.9 Randomization and Blinding

Enrolled participants will be assigned at random to one of two groups in a 1:1 ratio. Both study staff involved in evaluation of participants and participants are blinded to the assignments of participants to the study groups. We will conduct dynamic randomization so that it will be balanced by the following groups, in order of importance: anatomic site of lesion, HIV status, and time since diagnosis of the qualifying lesion (<12 months, ≥ 12 months). The qualifying lesion is defined as a histopathologically confirmed anal or vulvar HSIL diagnosed closest to, but on or after, 1/1/2014. Anatomic site will largely divide participants on gender, so further stratification by gender is unnecessary. Similarly, HIV status will be related to gender, as most women will be HIV negative while many men with anal HSIL (80% in our pilot study) will be HIV positive.

Please refer to the Randomization Standard Operating Procedure (SOP) for details about the randomization process for study staff involved in randomizing participants.

Randomization documentation and other pharmacy records will be stored in a secure location in the site pharmacy at each study location (VRC and UAB) apart from the rest of the participant file. This information will not be accessible to study staff members who

complete other study procedures with participants. Blinding will be maintained until all data are entered into the study database, all study endpoint data and other data included in the final analysis have been verified, and the data are ready for final analysis. If unblinding is needed for provision of medical treatment or to otherwise to protect the safety of study participants, DSMB input will be sought.

At the end of their study participation, individual participants will be offered the opportunity to be unblinded and provided their group assignment. Participants who received placebo will be offered the vaccine, free-of-charge.

## 5.10 Remote Consenting

Participants may be consented by telephone/telehealth as needed. The participant will speak with a qualified staff member to discuss study background, procedures, and any changes to the study (if re-consenting). Participants will have a chance to ask questions about all aspects of the study. Both the staff member and participant will have this discussion in private rooms. Prior to the discussion, the study staff member will confirm the participant's first and last name and date of birth.

The participant will be provided with a blank copy of the consent form. After the discussion is complete and all questions have been answered, the participant will sign the consent form and mail it to the clinic. The study staff member who conducted the discussion will sign the original consent form, make a copy of the fully executed consent form, and mail that copy to the participant. The original consent form will reside in a locked cabinet in the clinic. Written informed consent, HIPAA Authorization, and Medical Records and Tissue Releases will be obtained prior to participation or new procedures in the study.

## 5.11 Unblinding Participants

Due to the extension of the recruitment timeline, participants who entered the study early have been subjected to an extended waiting period to receive notification of their randomization assignment. The unblinding plan below provides an avenue to notify participants without compromising the blinded study design.

During the Month 42 phone call, participants will now be offered the opportunity to receive their randomization assignment. If a participant is not interested in receiving their assignment, they will not be unblinded until the end of the study. Participants confirming their interest in receiving their assignment will be contacted by unblinded study staff members and then will be notified of their assignment. Participants who received placebo will be offered the 9vHPV vaccine series free-of-charge. Those who accept will be scheduled for three vaccine visits scheduled at 0, 2, and 6 months. Only unblinded staff members will interact with unblinded participants, perform the vaccination visits, and have access to unblinded study documentation (e.g., unblinded case report forms, logs, schedules, etc.). The study team will not yet know the study results during the unblinding process.

At vaccination visits, a targeted physical exam will be performed as needed. Women of childbearing potential will undergo a urine pregnancy test prior to each vaccination.

The vaccine will be administered via intramuscular injection in the deltoid region of the preferred arm. Participants will be observed for 15 minutes after vaccine dose administration.

## 6 POTENTIAL RISKS & BENEFITS

#### 6.1 Potential Risks

<u>Phlebotomy</u>: Blood draw may cause faintness, discomfort and/or bruising. Rarely, an infection may develop.

Data Collection: Answering questions about medical history may be stressful.

<u>Pregnancy</u>: The safety of 9vHPV has not been established in pregnant women. Pregnant women will be excluded from the study at enrollment. Women who become pregnant will remain in the study and receive the remaining doses of the vaccine after the pregnancy resolves. Women who become pregnant after the 7<sup>th</sup> month of the study will remain in the study.

<u>Vaccination</u>: Safety of the vaccine after treatment for HSIL is unknown, but the vaccine is likely to be safe in this population. Since our study will result in off-label use, we will monitor safety by comparing type and frequency of AEs in the two study arms.

The most common adverse reaction in prior HPV trials was headache. Adverse reactions include fever, nausea, and dizziness; and local injection site reactions (pain, swelling, erythema, pruritus, and bruising). Syncope, sometimes associated with tonic-clonic movements and other seizure-like activity, has been reported following vaccination with 9vHPV and may result in falling with injury; observation for 15 minutes after administration is recommended. Anaphylaxis has been reported following vaccination with 9vHPV. As with any vaccination, there may be side effects that are not known at this time.

<u>Anal Swabs</u>: Putting a swab into the anus may cause some discomfort. Minor bleeding (less than a quarter of a teaspoon) rarely occurs in some people due to the insertion of the swabs. The bleeding stops almost immediately.

<u>High Resolution Anoscopy</u>: Insertion of an anoscope will likely cause some discomfort. Participants may feel pressure and the urge to have a bowel movement. Putting acetic acid (vinegar) in the anal canal rarely causes minor burning and irritation.

<u>Anal Biopsy</u>: Participants may have pain with the anal biopsies. Participants may have some bleeding for up to a week after biopsies, especially when they experience a bowel movement. There is a rare chance of very heavy bleeding that may require extra treatment. There is a very slight risk of infection (<1%). Participants will be instructed to contact the study clinic if they have symptoms of heavy bleeding or infection (fever, pain, redness, or swelling).

We will ask participants to refrain from receptive anal sex for 24 hours before the biopsy and to refrain from taking aspirin and ibuprofen, or medications containing these, prior to

the biopsy. This will help prevent any possible increase in risk of infection or bleeding after the procedure. We will instruct participants to avoid aggressive exercise immediately after the biopsy and to not engage in receptive anal sex one week after the rectal biopsy.

<u>Vulvoscopy</u>: Participants may feel discomfort during the procedure. Application of acetic acid for the exam may cause a burning sensation.

<u>Vulvar biopsy</u>: Injection of a local anesthetic prior to the biopsy maybe painful and the biopsy itself may cause pain, even with the use of an anesthetic. Biopsies may cause a pressure or tugging sensation. Bleeding and pain or irritation at the biopsy site(s) may continue for up to a week following the procedure. Although the skin biopsies are small (3-4mm), scarring may occur at the site. Participants will have to avoid sexual contact for 5 days after a biopsy, or until healing is complete.

<u>Lidocaine (injectable, +/- epinephrine)</u>: Lidocaine administration is associated with temporary pain and burning. Allergic reactions to lidocaine may occur, even in participants with no history of allergic reactions. Examples of allergic reactions include wheezing or difficulty in breathing, lightheadedness or fainting, skin rash and itching. As with any drug there may be unknown side effects. Biopsies may cause discomfort even when the area is numbed using lidocaine

<u>Silver nitrate</u>: Silver nitrate may be used if there is excessive bleeding after a biopsy. Allergic reactions to silver nitrate may occur, even in participants with no history of allergic reactions. Examples of allergic reactions include wheezing or difficulty in breathing, lightheadedness or fainting, skin rash and itching. As with any drug there may be unknown side effects.

<u>Monsel's Solution</u>: Topical Monsel's solution may be used for excessive bleeding after a rectal biopsy. There are no allergic reactions or adverse effects from application of Monsel's solution.

<u>Collection of Oral Rinse:</u> If a sample is collected when oral lesions are present, this may cause discomfort while using the oral mouthwash.

#### 6.2 Potential Benefits

Participants may benefit from the study by receiving the 9vHPV vaccine, otherwise, participants are not expected to benefit from participation in this trial. If this trial successfully shows that the HPV VLP vaccine is effective and provides proof for a conceptual framework, future studies could address immunogenicity over a longer time-period, and assess timing of doses with respect to HSIL diagnosis. If this trial shows that the HPV VLP vaccine is not a useful adjunctive care in this setting, future studies could determine if variant types in persistent infections or antibody assays could be employed as potential biomarkers of recurrence that could impact clinical surveillance.

#### 7 CLINICAL PROCEDURES

#### 7.1 Blood Collection

Blood will be obtained by routine venipuncture.

#### 7.2 HPV Swab Collection

Dacron swabs will be used to obtain a sample at the site of the qualifying lesion of the vulva or anus, depending on location of qualifying lesion for this study. Samples will be collected at Months 0, 18, 24, and 36.

For vulvar sampling, the swabs will be moved back and forth, in a tight zigzag motion from the clitoral prepuce down to the posterior fourchette, on one side and then the other, to allow collection on both sides of the perineum between the folds of the labia minora and majora.

Men and women with prior anal lesions will have a specimen collected by insertion of a dry swab 3–4 cm into the anal canal; the swab will be rotated once, and then removed with rotation and continued gentle pressure against the wall of the anal canal and perianal area.

Participants may choose to self-collect swabs of their qualifying lesion site for the Month 24 visit. If so, they will be instructed by study staff on how to collect the samples. However, all effort will be made for the swabs to be collected in-person by a study clinician.

Specimens will be placed in labeled collection tubes containing transport medium, the handle snapped off at the perforation, capped, and kept frozen at -20°C until assayed.

#### 7.3 HPV Oral Rinse Collection

For oral rinse sampling, participants will be asked to swish and deep gargle Scope solution for 30 seconds. The participant will spit the mouthwash into a specimen container. The specimen container will be capped, labeled, processed per SOP, and kept frozen at -20°C until assayed.

### 7.4 Data Collection

Participants will be asked questions about their health and anogenital pathology at the first and follow-up visits. Self-administered questionnaires will be completed at Enrollment, Month 6, Month 18, Month 24, and Month 36. Questions will focus on general health, medications, any new biopsies or surgeries, smoking history, sexual history, mental health, and daily activities. Report of any anogenital biopsies between study visits will trigger requests for pathology reports to review for anal or vulvar HSIL recurrences at the qualifying site.

We will retrieve medical records and pathology reports describing 1) treatment for AIN2/3-VIN2/3 (defined as the qualifying lesion, although the individual may have had other prior AIN2/3-VIN2/3 diagnoses prior to the qualifying diagnosis; and reports of 2) clinical and histopathological diagnosis of anal or vulvar HSIL that was done outside the study visits to

confirm recurrence of HSIL. The biopsies taken during follow up will be centrally reviewed by the study pathologist.

If HRA or vulvoscopy evaluation was done at a site other than the qualifying lesion, this information will be collected and will become part of the study record.

# 7.5 **High Resolution Anoscopy**

A digital anal/rectal exam will be performed. A lubricated plastic anoscope will be inserted into the anus. Then, a piece of gauze moistened with acetic acid is placed in the anus for 1-2 minutes to enhance visualization of abnormal areas. The anoscope will be put back into the anus. A colposcope is then used to visualize the skin inside the anus. Iodine may also be used to enhance visualization of lesions.

## 7.6 **Anal Biopsy**

The anal canal will be visualized during anoscopy. Topical lidocaine lubricant will be used to anesthetize the area, and lidocaine or bupivacaine may be injected if the lesion is near the anal verge on the perianal skin. A biopsy of an anal canal lesion is 2-3 mm.

## 7.7 Vulvoscopy

In dorsal lithotomy position, the entire vulva, mons, and perianal area will be inspected for lesions. Acetic acid will be applied liberally to the entire area for 3-5 minutes. Careful examination will be performed with a colposcope and any suspicious lesions will be identified by location and clinical impression.

# 7.8 **Vulvar Biopsy**

The vulva will be prepped with chlorhexidine or Betadine solution. Approximately 1cc of 1% lidocaine (+/- epinephrine) will be injected to anesthetize the area for biopsy. 3 or 4 mm punch biopsy will be used to take biopsy. Silver nitrate may be used as a cautery agent to control bleeding.

#### 8 LABORATORY PROCEDURES

Laboratory procedures include HIV testing, HPV DNA typing and variant sequencing, and HPV serology. Centralized pathology review of qualifying lesion tissue samples and potential recurrences will be reviewed at the UW (by Dr. V. Grieco). Future studies using samples collected in this study will need to be approved by the Institutional Review Board.

Assays may also be conducted with researchers from other universities and from pharmaceutical companies.

# 8.1 Urine Pregnancy Testing

Urine pregnancy testing will be performed per manufacturer's guidelines.

## 8.2 HIV-1 Antibody Testing

HIV-1 antibody testing will be performed at Screening Visit, as needed. HIV-1 testing will be repeated if previous testing was performed > 12 months prior to the Screening visit (> 6 months for high risk participants).

# 8.3 HPV Capsid Antibody Analysis

Serum will be drawn into a red-top tube, processed and delivered to the laboratory for HPV capsid antibody assays.

# 8.4 HPV Typing from Tissue

Investigators will retrieve tissue associated with the qualifying lesion and recurrent diagnoses from study clinicians or, if between visits, local providers. All tissue blocks will be reviewed and sectioned for HPV DNA testing by Dr. Grieco. We will perform HPV typing and HPV16 lineage assessment on HPV16 positive samples.

# 8.5 **HPV Typing from Oral Samples**

Oral rinse specimens will be collected at Screening, and Months 7, 18, 24, and 36 for type-specific HPV using polymerase chain reaction (PCR)-based method according to the protocol recommended by the manufacturer.

#### 8.6 Future Genetic Research

Samples will be collected for future genetic studies of HPV-related conditions using DNA from blood collected at Month 7. All such studies will be performed by the study Investigators or their scientific collaborators and will be reviewed and approved by the Institutional Review Board.

#### 9 STUDY PRODUCT

#### 9.1 **Treatment Groups**

| Name | Dose | How administered |
|---|---|---|
| Gardasil® | 0.5 ml dose | Intramuscular injection in the deltoid region of the arm |
| Placebo | 0.5 ml saline | Intramuscular injection in the deltoid region of the arm |

## 9.2 Study Product and Source

Gardasil: Pre-filled vials with vaccine (Gardasil, 9vHPV) will be obtained from Merck. The 9vHPV vaccine is FDA approved.

Placebo: Normal saline will be obtained from a commercial manufacturer.

## 9.3 Storage

9vHPV: The vaccine will be stored at 2 to 8°C (36 to 46°F) and protected from light until use. The vaccine will be administered as soon as possible after being removed from refrigeration.

Placebo: The placebo will be stored per package guidelines.

#### 9.4 Recommended Dose and Schedule

Each 0.5-mL dose of 9vHPV contains approximately 30 mcg of HPV Type 6 L1 protein, 40 mcg of HPV Type 11 L1 protein, 60 mcg of HPV Type 16 L1 protein, 40 mcg of HPV Type 18 L1 protein, 20 mcg of HPV Type 31 L1 protein, 20 mcg of HPV Type 33 L1 protein, 20 mcg of HPV Type 45 L1 protein, 20 mcg of HPV Type 52 L1 protein, and 20 mcg of HPV Type 58 L1 protein. Each 0.5-mL dose of the vaccine also contains approximately 500 mcg of aluminum (provided as AAHS), 9.56 mg of sodium chloride, 0.78 mg of L-histidine, 50 mcg of polysorbate 80, 35 mcg of sodium borate. The product does not contain a preservative or antibiotics.

Participants will be administered vaccine at 0, 2, and 6 months, as per the 9vHPV package insert. The preferred injection site is the deltoid muscle, preferably in the non-dominant arm, with intramuscular deposition.

#### 9.5 Administration

9vHPV should be thoroughly shaken before use and administered as soon as possible after being removed from refrigeration. After thorough agitation, 9vHPV is a white, cloudy liquid. Parenteral drug products should be inspected visually for particulate matter and discoloration prior to administration. The product should not be used if particulates are present or if it appears discolored.

The placebo (0.5 ml saline) will be prepared by the site pharmacist or clinician per package guidelines.

All participants will be observed for syncope for 15 minutes after vaccine dose administration, as syncope has been reported following vaccination with 9vHPV. The CDC Vaccine Information Sheet will be given with each vaccination to the participant.

## 9.6 Contraindications

Hypersensitivity, including severe allergic reactions to yeast (a vaccine component).

# 9.7 **Blinding**

An unblinded research pharmacist or clinician will administer the immunization to maintain the blind, as per clinic standard procedures.

## 9.8 Study Product Accountability

The research staff will maintain complete records of all study products received and subsequently dispensed.

#### 10 ASSESSMENT OF SAFETY

#### 10.1 Adverse Events

The investigator is responsible for reporting Adverse Events (AEs) that are observed or reported during the study.

#### 10.2 **Definition of Adverse Event**

An adverse event (AE) is defined as any untoward medical occurrence in a participant including any abnormal sign (e.g., abnormal physical exam), symptom, or disease, temporally associated with the subject's participation in the research, which does not necessarily have a causal relationship with the study. Mechanisms of obtaining information on AE will rely primarily on visits to the clinic with a health care provider.

The occurrence and severity of all AEs will be listed and graded according to the FDA criteria (FDA Guidance for Industry: Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials). The following information will be collected on all AEs experienced during this study:

- Name of the event: If the event is described in the FDA Toxicity Grading Scale, the Investigator should use that terminology. Otherwise, terminology that clearly describes the pathophysiology of the event and body system affected should be used.
- Onset Date
- Date of resolution
- Severity
  - If an event is not described in the FDA Toxicity Grading Scale and therefore not graded, the following grading will be used:
    - 1. Mild, easily tolerated by the participant, causing minimal discomfort and not interfering with everyday activities.
    - 2. Moderate, sufficiently discomforting to interfere with normal everyday activities
    - 3. Severe, prevents normal everyday activities
    - 4. Life-threatening, places the participant at immediate risk for death
- Relationship to study drug: All AEs will have a causality assessment performed at the time of reporting the event to document the Investigator's perception of causality.
   For the purposes of this study, causality will be assigned using the following criteria:

- Related: The event cannot be attributed to the participant's underlying medical condition or other concomitant therapy and there is a compelling temporal association between the onset of the events and study drug administration that leads the Investigator to believe that there is reasonable chance of a causal relationship.
- o Remote: A relationship is not obvious but cannot be ruled out.
- Not related: The participant's underlying medical condition or concomitant therapy can easily be identified as the cause of the event and there is no temporal relationship between the event and the study drug.

# 10.3 Definition of Serious Adverse Event (SAE)

The Investigator is required to determine if each AE was an SAE. An SAE is any AE occurring at any administration of study drug that results in any of the following outcomes:

- Death
- A life-threatening adverse drug experience
- A congenital anomaly or birth defect
- Inpatient hospitalization (hospitalizations for elective medical/surgical procedures, scheduled treatments, or routine check-ups are not SAE by these criteria)
- A persistent or significant disability / incapacity

Important medical events that may not meet any of the above criteria may be considered an SAE when, based upon appropriate medical judgment, it may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed above.

#### 10.4 Adverse Event Reporting

The following AEs will be collected during the study on appropriate source documentation:

- Vaccine-related AEs will be collected
- Reactogenicity will be collected though Day 5 after each dose.
- Biopsy-related AEs will be collected until healing after each biopsy.
- SAEs will be recorded until the final study visit.

Adverse Events that will be recorded in the study database are reactogenicity and any Grade 3 or higher AEs that are deemed related or possibly related to the study. All Serious Adverse Events (SAEs) will be recorded.

Please refer to the AE Documentation Standard Operating Procedure (SOP) for details about the AE documentation for study staff involved in clinical evaluation of the participants.

Information to be collected includes event description, date of onset, investigator assessment of severity, investigator assessment of relationship to study product, date of resolution of the event, seriousness, and outcome. The **intensity** of nonserious AEs can be assessed by a licensed clinician (i.e., physician, nurse, Nurse Practitioner, Physician Assistant). **Causality** of nonserious AEs can be assessed only by a clinician licensed to

make medical diagnoses (ie, physician, Nurse Practitioner, Physician Assistant). All AEs will be followed to adequate resolution or until considered stable.

Any medical condition that is present at screening will be considered as baseline and will not be reported as an AE. If the severity of any pre-existing medical condition increases during the study period, then it will be recorded as an AE.

# 10.4.1 **SAE Reporting**

All SAEs will be reported immediately to Dr. Wald at either site and also to Dr. Huh if at UAB.

The UAB 24-hour emergency number is 205-934-3411.

SAE Alternate: A clinician from the Virology Research Clinic is available at any time by calling the 24-hour emergency pager at 206-598-0924 and asking for the Virology Research Clinic Clinician on-call.

All SAEs will be recorded on the appropriate SAE Report Form. The SAE report will include the following information (as available):

- Participant ID
- Description of SAE (onset date, severity, causal relationship)
- Basic demographic information
- Outcomes attributed to the event
- Summary of relevant test results, laboratory data, and other relevant history
- The first and last dates of study drug administration
- Statement of whether study drug was discontinued or schedule modified
- Statement of whether the event abated after study drug was discontinued or schedule modified
- Statement of whether the event recurred after reintroduction of the study drug if it had been discontinued.

All SAEs reported will be relayed to the Human Subjects Division (HSD) of the University of Washington as required by HSD policy.

# 10.4.2 Follow-up of SAE

All SAEs will be followed through resolution by a study physician.

## 10.5 Safety Monitoring

## 10.5.1 Data and Safety Monitoring Plan

Institutional support of trial monitoring will be in accordance with the FHCRC/University of Washington Cancer Consortium Institutional Data and Safety Monitoring Plan. Under the provisions of this plan, FHCRC Clinical Research Support (CRS) coordinates data and compliance monitoring conducted by consultants, contract research organizations, or FHCRC employees unaffiliated with the conduct of the study. Independent monitoring

visits occur at specified intervals determined by the assessed risk level of the study and the findings of previous visits per the institutional DSMP.

In addition, protocols are reviewed at least annually and as needed by the Consortium Data and Safety Monitoring Committee (DSMC), FHCRC Scientific Review Committee (SRC) and the FHCRC/University of Washington Cancer Consortium Institutional Review Board (IRB). The review committees evaluate accrual, adverse events, stopping rules, and adherence to the applicable data and safety monitoring plan for studies actively enrolling or treating subjects. The IRB reviews the study progress and safety information to assess continued acceptability of the risk-benefit ratio for human subjects. Approval of committees as applicable is necessary to continue the study.

The trial will comply with the standard guidelines set forth by these regulatory committees and other institutional, state and federal guidelines.

## 10.5.2 Data and Safety Monitoring Board

We will convene a Data Safety Monitoring Board (DSMB) for this study. DSMB members will be recruited from among HPV vaccine and oncology experts in the Seattle area (chair and 3 members); one of the four members will be the lead biostatistician for the trial and the biostatistician for the DSMB, Amalia Magaret, PhD and there will also be an independent statistician participating. Prior to any participant enrollment in the study, DMSB members will form an understanding of the protocol and definitions being used, and review and approve the charter.

The DSMB will conduct two independent reviews of the interim safety data, the first after the initial 50 participants complete two immunizations and the second after 150 participants complete their Month 6 Visit. In addition, any grade 3 or higher AEs that occur in more than 10% of the participants, except for local and systemic immunogenicity, will be reviewed by the DSMB chair who will then consult the remaining members. The DSMB will review data upon their request as specified in the charter.

#### 11 CLINICAL MANAGEMENT

The clinic visits for this study will be conducted over a 36-month period for each participant. During this period, participants will be seen at clinic for injections, surveillance and study sample collection. Participants will be asked to complete one final phone call visit at Month 42.

Participants who opted to be unblinded at the end of their participation (Month 42), received placebo, and chose to receive the 9vHPV vaccine, will return to the research clinic at 0, 2, and 6 months for vaccination.

## 11.1 Participant Withdrawal or Discontinuation

Normal study completion will be defined as completion of the 36-months of clinic visits plus an additional telephone interview at 42 months (or mid-point between the end of the

clinic visits and the end of data collection for the study). Participants who do not appear for scheduled visits will be traced using originally provided contact information. Efforts will be made to accommodate participants who are willing to return to clinic outside of scheduled visit windows in order to maximize ascertainment.

Participants may voluntarily withdraw from the study for any reason at any time. The investigators may also withdraw participants from the study at any time to protect patient safety, if the patient is unwilling or unable to comply with required study procedures, for administrative reasons, at the request of government or regulatory agencies, or if the study is terminated early. Study staff members will record the reason(s) for withdrawal in participants' study records.

#### 12 DATA MANAGEMENT

#### 12.1 Data Collection

Data collection will involve questionnaires, specimen collection, and results of laboratory testing that are obtained specifically for research purposes. All participants are tracked though a unique study identification number. This number is the only unique identifier that will appear on the participant questionnaires, specimens and the databases into which these data will be entered.

Research records for participants in this study are the responsibility of the investigators. All study documents will be confidential.

Tracking data, which contains PHI, is password protected and stored on secure servers. Paper files, such as interviewer contact sheets with PHI and study identifiers, are stored separately in locked file cabinets when not in use at the VRC or UAB.

## 12.2 Case Report Forms (CRF)

Case Report Forms will be identified with a study number. CRFs are to be completed for each participant by the investigator or designated member of the study staff and initialed by the investigator or designee. CRFs will be completed neatly and legibly. Any modification of previously entered data must be made by the investigator or designee by striking through the original entry with a single line, initialing and dating changes, and entering the correct data nearby. A valid explanation must be given for any missing information. All data will be entered into a computer database and a further quality control check will be made to produce a final database for analysis.

#### 13 HUMAN SUBJECTS PROTECTIONS

## 13.1 IRB Approval

Prior to the initiation of the study, the principal investigator will obtain written approval to conduct the study from the University of Washington Human Subjects Review Committee.

## 13.2 Informed Consent

The investigator or study coordinator will explain the purpose and nature of the study, including potential benefits and risks to the participant, to each potential participant before enrollment in the study. Non-English readers will be consented using the short-form consent process with a qualified interpreter.

The participant must sign an informed consent form approved by the IRB before entering the study. All original informed consent forms will be retained by the Principal Investigator separately from the participant's records, as they have names. The participant will receive a copy of the signed informed consent form.

# 13.3 Protection against Risk

All procedures are conducted in a clinical setting with experienced research clinicians and coordinators. Information and samples are coded to protect the confidentiality of the participants and no identifying information of any kind is released to any other person or agency without specific written permission. Only the clinic staff will have access to potentially identifiable personal information. All research staff is skilled at maintaining confidentiality of the participants and their study results. All data are coded and files are maintained in locked cabinets.

We have established Standard Operating Procedures to minimize the risk of study procedures. Care will be taken during the consenting process and throughout the study to assure that participants are fully informed of all study procedures and associated risks. Participants will also be educated about how to contact the study investigators if any questions or concerns arise.

#### 14 STUDY DESIGN DETAILS

## 14.1 Sample size

For the virologic primary aim, 212 patients are required to have a 90% chance of detecting, as significant at the 5% level, a decrease in the primary outcome measure, persistent high-risk, vaccine-type infection, of 50%, from approximately 40% in the control group to 20% in the experimental group. The 50% reduction is based on prior studies of the impact of 4vHPV on recurrence<sup>6, 18</sup> and the prevalence of approximately 40% hrHPV in HSIL treated controls during long-term follow up.<sup>19</sup> We anticipate that with 4% dropout, we will need to enroll approximately 230 participants to meet the primary aim.

#### 14.2 Randomization

Participants will be randomized 1:1 to receive vaccine or placebo as equal randomization is the most efficient approach to trial design as it minimizes sample size and maximizes information obtained on both arms.<sup>19</sup> See Section 5.8 for details of randomization.

## 15 STATISTICAL CONSIDERATIONS

## 15.1 Missing data and loss to follow-up

As mentioned above, we will enroll 21 additional participants so that if 10% of our planned cohort does not complete 3 years of recurrence assessments, we will still be powered to detect our aims of interest. Nonetheless, as described in the protocol, efforts will be made to contact participants who do not appear for scheduled visits, and they will be encouraged to continue their study commitment. Loss to follow-up will be monitored and compared between arms, and reasons for discontinuation will be recorded, if available. We will measure potential differential follow-up by vaccination status, and the potential for loss to follow-up to be associated with the study outcome (either those with recurrence are more likely or less likely to attend). Methods for evaluation of the primary aim may differ depending on whether differential follow-up is observed.

#### 15.2 Visit Windows

Participants will have swabs and oral rinses for HPV detection at 0, 18, 24, and 36 months, and undergo surveillance for HSIL at 0, 18 and 36 months, using visualization via anoscopy or vulvoscopy, with a biopsy if a lesion is detected. As recurrences are anticipated to be detected early by study surveillance, it is unlikely that participants will present for earlier diagnosis between scheduled visits, but information on HSIL diagnosed outside the study will be collected from medical records. In analysis, we will use timing of detection of the recurrence rather than imputing the possible timing of recurrence itself. While the time between visit windows is 18 months, comparison of survival-type and cumulative incidence type sample size calculations demonstrate that obtaining the timing of event is not critical to determining a difference in hazard of event by arm. With annual incidence of recurrence  $\lambda_C$  = 12%, the median time to recurrence is -ln(1-.5)/.12 = 5.8 years. On the vaccine it will take twice as long, 11.7 years. These large differences do not require short visit windows to detect persistent infection or recurrences.

# 16 STATISTICAL ANALYSIS PLAN

## 16.1 Data handling

We anticipate some participants will miss visits, which adds uncertainty to the timing of events. For those who have a high-risk persistent infection or a recurrence detected following a missed visit(s), a sensitivity analysis will be performed setting the timing of the recurrence first to its detection date and secondly to the date of that earliest missed visit prior to detection. Other violations, such as failure to complete all vaccine doses, will be handled by comparison of the Intention to Treat (ITT) and Per Protocol (PP) analyses.

#### 16.2 Analysis populations

The ITT population will be those enrolled and randomized and for whom events accrue starting at day 30 after the first dose of the vaccine. The PP population will be those who completed all phases of vaccine and did not have a subsequent HSIL within 1 month of the last dose. Efficacy analyses will be conducted on both the ITT and PP populations, with the ITT population considered primary. The safety population is the same as the ITT population.

# 16.3 Primary endpoint

We will evaluate vaccine efficacy against persistent 9vHPV hrHPV infection detected between months 18 and 36. Persistence will be measured as two or more consecutive PCR positive swabs for the same HPV genotype. We will use Cox proportional hazards to compare time start of interval for the persistent infection in the vaccinated to unvaccinated group.

In secondary analyses we will adjust for factors upon which participants were stratified: anatomic site, HIV status (positive vs negative), time since diagnosis (<12 months, >12 months). We will also assess balance with regard to smoking status and include it in secondary models. We will assess whether to include smoking as a binary covariate, and we will assess using current consumption levels among smokers. Graphical depictions of endpoint rates by levels of smoking can help determine appropriate parameterization.

## 16.4 Secondary endpoints

Secondary analyses will include additional exposures or on subsets.

#### Sub-Aim 1.

For Sub-Aim 1, we will evaluate differences in the hazard of recurrence using Cox proportional hazards in the ITT population and the PP population, if appropriate; see contingencies for departures from model assumptions below. As this is a randomized trial, the primary analysis will include no other potential predictors of recurrence except for the treatment arm: vaccine *vs.* placebo. However, additional known risk factors will be included in secondary analyses of the primary aim, to confirm findings and to adjust for potential imbalances that occurred during randomization.

## Sub-Aim 2.

We will divide the study data by treatment arm in order to assess Sub-Aim 2, evaluating placebo and vaccine recipients separately. We will assess whether presence and amount of HPV antibody, detected at baseline in the placebo arm, is protective against recurrence. Subsequent graphical analysis examining incidence of recurrence by quartiles and deciles of antibody level will allow visual assessment of the relationship between levels of antibody and risk of recurrence. In further exploratory analyses for this sub-Aim, for the vaccine arm, we will assess whether magnitude of vaccine antibody levels month 1 following the third vaccination in the vaccine arm affects recurrence. Should a cutoff be observed, we may be able to determine the level of antibody (by titer) associated with protection.

#### Sub-Aim 3.

We will evaluate vaccine efficacy against persistent 9vHPV hrHPV oral infection detected between months 18 and 36. Persistence will be measured as two or more consecutive PCR positive swabs for the same HPV genotype from oral samples. We will use Cox proportional hazards to compare time start of interval for the persistent infection in the vaccinated to unvaccinated groups.

#### 16.5 Departures from model assumptions

If the hazards of recurrence by arm are not proportional but do not cross, a log rank test is most powerful to detect the alternative hypothesis of vaccine benefit. However, should the hazards appear to cross, we will make use of current powerful methods, such as those suggested by Liu or Li.<sup>20,21</sup> If informative censoring is suspected, alternative analytical

methods may be employed such as a recent one by Zhao which address informative censoring through imputation, without modeling the underlying censoring mechanism.<sup>22</sup>

## 16.6 Left truncation

Some persons will not be eligible for inclusion in per-protocol analysis of the primary or first secondary aim because their recurrence occurs prior to 1 month post third vaccination. This affects persons in both arms in a placebo-controlled trial. Should the vaccine be partially effective after only one or two doses, there may be a smaller number of persons recurring during the vaccination series in the active vaccine arm versus the placebo arm. Comparison of the included populations and of the results between the ITT and PP analyses will help elucidate this possibility.

## 17 REFERENCES

- Saraiya M, Unger ER, Thompson TD, Lynch CF, Hernandez BY, Lyu CW, Steinau M, Watson M, Wilkinson EJ, Hopenhayn C, Copeland G, Cozen W, et al. US Assessment of HPV Types in Cancers: Implications for Current and 9-Valent HPV Vaccines. *J Natl Cancer Inst* 2015;107.
- 2. Stier EA, Abbasi W, Agyemang AF, Valle Álvarez EA, Chiao EY, Deshmukh AA. Brief Report: Recurrence of Anal High-Grade Squamous Intraepithelial Lesions Among Women Living With HIV. *Jaids-J Acq Imm Def* 2020;**84**: 66-9.
- 3. Jones RW, Rowan DM, Stewart AW. Vulvar intraepithelial neoplasia: aspects of the natural history and outcome in 405 women. *Obstet Gynecol* 2005;**106**: 1319-26.
- 4. Carter JJ, Madeleine MM, Shera K, Schwartz SM, Cushing-Haugen KL, Wipf GC, Porter P, Daling JR, McDougall JK, Galloway DA. Human papillomavirus 16 and 18 L1 serology compared across anogenital cancer sites. *Cancer Res* 2001;61: 1934-40.
- 5. Miltz A, Price H, Shahmanesh M, Copas A, Gilson R. Systematic Review and Meta-Analysis of L1-VLP-Based Human Papillomavirus Vaccine Efficacy against Anogenital Pre-Cancer in Women with Evidence of Prior HPV Exposure. *PLoS One* 2014;**9**: e90348.
- 6. Swedish KA, Factor SH, Goldstone SE. Prevention of recurrent high-grade anal neoplasia with quadrivalent human papillomavirus vaccination of men who have sex with men: a nonconcurrent cohort study. *Clin Infect Dis* 2012;**54**: 891-8.
- 7. Kang WD, Choi HS, Kim SM. Is vaccination with quadrivalent HPV vaccine after loop electrosurgical excision procedure effective in preventing recurrence in patients with high-grade cervical intraepithelial neoplasia (CIN2-3)? *Gynecol Oncol* 2013;**130**: 264-8.
- 8. Wilkin TJ, Chen H, Cespedes MS, Leon-Cruz JT, Godfrey C, Chiao EY, Bastow B, Webster-Cyriaque J, Feng Q, Dragavon J, Coombs RW, Presti RM, et al. A randomized, placebo-controlled trial of the quadrivalent HPV vaccine in HIV-infected adults age 27 years or older: AIDS Clinical Trials Group protocol A5298. *Clin Infect Dis* 2018;**67**: 1339-46.
- 9. WHO, Weekly Epidemiological Record, 24 October 2014. Human papillomavirus vaccines: WHO position paper, October 2014, 2014.
- 10. IARC, Primary End-points for Prophylactic HPV Vaccine Trials, IARC Working Group Report, Vol. 7, 2014.
- 11. Rositch AF, Koshiol J, Hudgens MG, Razzaghi H, Backes DM, Pimenta JM, Franco EL, Poole C, Smith JS. Patterns of persistent genital human papillomavirus infection among women worldwide: A literature review and meta-analysis. *International Journal of Cancer* 2013;**133**: 1271-85.
- 12. Vaccarella S, Söderlund-Strand A, Franceschi S, Plummer M, Dillner J. Patterns of human papillomavirus types in multiple infections: an analysis in women and men of the high throughput human papillomavirus monitoring study. *PLoS One* 2013;8: e71617.

- 13. Joura EA, Giuliano AR, Iversen OE, Bouchard C, Mao C, Mehlsen J, Moreira ED, Jr., Ngan Y, Petersen LK, Lazcano-Ponce E, Pitisuttithum P, Restrepo JA, et al. A 9-Valent HPV Vaccine against Infection and Intraepithelial Neoplasia in Women. *N Engl J Med* 2015;**372**: 711-23.
- 14. Castellsague X, Giuliano AR, Goldstone S, Guevara A, Mogensen O, Palefsky JM, Group T, Shields C, Liu K, Maansson R, Luxembourg A, Kaplan SS. Immunogenicity and safety of the 9-valent HPV vaccine in men. *Vaccine* 2015;**33**: 6892-901.
- 15. Van Damme P, Olsson SE, Block S, Castellsague X, Gray GE, Herrera T, Huang LM, Kim DS, Pitisuttithum P, Chen J, Christiano S, Maansson R, et al. Immunogenicity and Safety of a 9-Valent HPV Vaccine. *Pediatrics* 2015;**136**: e28-e39.
- 16. Kahn JA, Xu J, Kapogiannis BG, Rudy B, Gonin R, Liu N, Wilson CM, Worrell C, Squires KE. Immunogenicity and safety of the human papillomavirus 6, 11, 16, 18 vaccine in HIV-infected young women. Clin Infect Dis 2013;57: 735-44.
- 17. Slade BA, Leidel L, Vellozzi C, Woo EJ, Hua W, Sutherland A, Izurieta HS, Ball R, Miller N, Braun MM, Markowitz LE, Iskander J. Postlicensure safety surveillance for quadrivalent human papillomavirus recombinant vaccine. *JAMA* 2009;**302**: 750-7.
- 18. Joura EA, Garland SM, Paavonen J, Ferris DG, Perez G, Ault KA, Huh WK, Sings HL, James MK, Haupt RM. Effect of the human papillomavirus (HPV) quadrivalent vaccine in a subgroup of women with cervical and vulvar disease: retrospective pooled analysis of trial data. *BMJ* 2012;**344**: e1401.
- 19. Frega A, Sopracordevole F, Scirpa P, Biamonti A, Lorenzon L, Scarani S, De SL, Pacchiarotti A, Moscarini M, French D. The re-infection rate of high-risk HPV and the recurrence rate of vulvar intraepithelial neoplasia (VIN) usual type after surgical treatment. *Med Sci Monit* 2011;**17**: CR532-CR5.
- 20. Liu K, Qiu P, Sheng J. Comparing two crossing hazard rates by Cox proportional hazards modelling. *Stat Med* 2007;**26**: 375-91.
- 21. Li H, Han D, Hou Y, Chen H, Chen Z. Statistical inference methods for two crossing survival curves: a comparison of methods. *PLoS One* 2015;**10**: e0116774.
- 22. Zhao Y, Herring AH, Zhou H, Ali MW, Koch GG. A multiple imputation method for sensitivity analyses of time-to-event data with possibly informative censoring. *Journal of biopharmaceutical statistics* 2014;**24**: 229-53.

#### **APPENDIX A: STUDY VISIT WINDOWS**

# VIVA Visit Windows \*\*Month defined as 30 days

| Visit | STUDY MONTH | ORIGINAL VIST WINDOW | COVID-ADJUSTED<br>VISIT WINDOWS* |
|---|---|---|---|
| 0 | Screening | | |
| 1 | Enrollment/Month 0 (Dose 1) | Within 56 days of screen | |
| 2 | Month 2 Visit (Dose 2) <sup>1</sup> | at least 28 days from Dose 1 | |
| 3 | Month 6 Visit (Dose 3) <sup>2</sup> | at least 3 months from Dose 2 AND At least 5 months from Dose 1 | |
| 4 | Month 7 Visit <sup>3</sup> | + 14 days | + 30 days |
| 5 | Month 12 Visit (phone) | - 60 / + 90 days | - 60 / + 120 days |
| 6 | Month 18 Visit | - 60 / + 90 days | - 60 / + 120 days |
| 7 | Month 24 Visit | - 60 / + 90 days | - 60 / + 120 days |
| 8 | Month 36 Visit | - 60 / + 90 days | - 60 / + 120 days |
| 9 | Month 42 Visit (phone) | - 60 / + 90 days | - 60 / + 120 days |

<sup>&</sup>lt;sup>1</sup> Dose 2 can be given at a maximum allowable time of 9 months post Dose 1

### References:

https://www.cdc.gov/mmwr/preview/mmwrhtml/rr6305a1.htm http://www.immunize.org/askexperts/experts hpv.asp

The minimum interval between the first and second doses of vaccine is 4 weeks. The minimum interval between the second and third doses of vaccine is 12 weeks. The minimum interval between the first and third doses is 5 calendar months. If the vaccination series is interrupted, the series does not need to be restarted.

<sup>&</sup>lt;sup>2</sup> Dose 3 can be given at a maximum allowable time of 12 months post Dose 1.

<sup>&</sup>lt;sup>3</sup> The Month 7 Visit is targeted for 1 month after Dose 3.

<sup>\*</sup>Due to the COVID-19 outbreak, the maximum allowable times and window dates will be relaxed for participants whose visit schedules were affected due to clinic closures and/or restrictions.

**APPENDIX B: TABLE OF PROCEDURES** 

| | | | | | | Study | Mont | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | Screen<br>(-1) | Enrollment (Month 0) | nt | 12 | 18 | 24 | 36 | 42 | | |
| Obtain Informed Consent | Х | | | | | | | | | |
| Review Inclusion/Exclusion<br>Criteria | Х | Х | | | | | | | | |
| Medical History and PE | Х | | | | | | | | | |
| Interim History and Targeted PE | | Х | Х | Х | Х | | Х | Х | Х | |
| HIV Testing (as needed) | Х | | | | | | | | | |
| Urine Pregnancy Test (women only) | Х | Х | Х | Х | | | | | | |
| Randomization | | Х | | | | | | | | |
| Vaccination | | Х | Х | Х | | | | | | |
| Self-Administered Questionnaire | | Х | | Х | | | Х | Х | Х | |
| Blood Draw - Serum (up to 20 cc) | | Х | | | Х | | Х | | Х | |
| Blood Draw for DNA (optional) | | | | | Х | | | | | |
| Oral Rinse | Х | | | | Х | | Х | Х | Х | |
| Anoscopy/Vulvoscopy | X <sup>2</sup> | | | | | | Х | | Х | |
| Swab for HPV | Х | | | | | | Х | <b>X</b> <sup>5</sup> | Х | |
| Biopsy | X <sup>3</sup> | | | | | | <b>X</b> <sup>3</sup> | | X <sup>3, 4</sup> | |
| Telephone Visit | | | | | | Х | | | | Х |

<sup>&</sup>lt;sup>1</sup>Reminder calls will be conducted every 1-3 months after the Month 7 visit for study retention.

<sup>&</sup>lt;sup>2</sup> Anoscopy/vulvoscpy will not be performed if the procedure was done within 8 weeks of the Screening Visit with clinical co-Investigators or an ANCHOR-certified provider.

<sup>&</sup>lt;sup>3</sup> Biopsy, as needed, if lesion is noted at qualifying site during anoscopy/vulvoscopy

<sup>&</sup>lt;sup>4</sup> If no lesion indicating a biopsy is needed is visible, an optional biopsy will be performed at the site of qualifying lesion.

<sup>&</sup>lt;sup>5</sup> Swab collection may be done by either a study clinician or self-collected.

<sup>&</sup>lt;sup>6</sup>Participants who opted to be unblinded at the end of their participation (Month 42), received placebo, and chose to receive the 9vHPV vaccine, will return to the research clinic at 0, 2, and 6 months for vaccination with the 9vHPV vaccine free-of-charge.